CLINICAL TRIAL: NCT00876395
Title: A Randomized Phase III, Double-Blind, Placebo-Controlled Multicenter Trial of Everolimus in Combination With Trastuzumab and Paclitaxel, as First Line Therapy in Women With HER2 Positive Locally Advanced or Metastatic Breast Cancer
Brief Title: Everolimus in Combination With Trastuzumab and Paclitaxel in the Treatment of HER2 Positive Locally Advanced or Metastatic Breast Cancer
Acronym: BOLERO-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001J2301; 2008-006556-21 (EudraCT Number)
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; HER2+; mTOR; everolimus; RAD001; first line; metastatic; locally advanced; Trastuzumab; Paclitaxel; First Line Therapy; HER2 Positive; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Everolimus; Trastuzumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Everolimus + Paclitaxel + Trastuzumab (Experimental): Everolimus 10 mg daily in combination with paclitaxel 80mg/m2 weekly on days 1, 8, 15 and trastuzumab 2mg/kg weekly on days 1, 8, 15, 22
  Interventions: Drug: Everolimus; Drug: Trastuzumab; Drug: Paclitaxel
- Placebo + Paclitaxel + Trastuzumab (Placebo Comparator): Placebo of everolimus 10 mg daily in combination with paclitaxel 80mg/m2 weekly on days 1, 8, 15 and trastuzumab 2mg/kg weekly on days 1, 8, 15, 22
  Interventions: Drug: Placebo; Drug: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Everolimus — Everolimus was administered in a continuous oral daily dosing of 10 mg (two 5-mg tablets).
  Other Names: RAD001
  Arms: Everolimus + Paclitaxel + Trastuzumab
Drug: Placebo — Everolimus placebo was administered in a continuous oral daily dosing of 10 mg (two 5-mg tablets).
  Arms: Placebo + Paclitaxel + Trastuzumab
Drug: Trastuzumab — Trastuzumab, 2 mg/kg weekly was used intravenously.
Drug: Paclitaxel — Paclitaxel, 80 mg/m2 weekly was used intravenously.

SUMMARY:
The purpose of this Phase III study was to confirm the value of adding everolimus to weekly paclitaxel and trastuzumab as treatment of HER2-overexpressing metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult Women (≥ 18 years old).
* Histologically or cytologically confirmed invasive breast carcinoma with local recurrence or radiological evidence of metastatic disease.
* Must have at least one lesion that can be accurately measured or bone lesions in the absence of measurable disease.
* HER2+ patients by local laboratory testing (IHC 3+ staining or in situ hybridization positive).
* Prior trastuzumab and/or chemotherapy (taxanes included) as neo-adjuvant or adjuvant treatment is allowed but should be discontinued > 12 months prior to randomization.
* Prior treatment for breast cancer with endocrine therapy (adjuvant or metastatic settings) is allowed but should be discontinued at randomization. Patients treated with bisphosphonates at entry or who start bisphosphonates during study may continue this therapy during protocol treatment.
* Documentation of negative pregnancy test.
* Organ functions at time of inclusion.

Exclusion Criteria:

* Prior mTOR inhibitors for the treatment of cancer.
* Other anticancer therapy for locally advanced or metastatic breast cancer except for prior hormonal therapy.
* Patients with only non-measurable lesions other than bone metastasis (e.g. pleural effusion, ascites, etc).
* Radiotherapy to ≥ 25% of the bone marrow within 4 weeks prior to randomization
* History of central nervous system metastasis.
* Impairment of gastrointestinal (GI) function or GI disease or active ulceration of the upper gastrointestinal tract.
* Serious peripheral neuropathy.
* Cardiac disease or dysfunction.
* Uncontrolled hypertension.
* HIV.
* Pregnant,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2009-09-10 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (129):
- United States (25):
  - University of South Alabama / Mitchell Cancer Institute Dept. of Mitchell Cancer Inst., Mobile, Alabama
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Comprehensive Blood and Cancer Center Dept. of CBCC (2), Bakersfield, California
  - St. Jude Heritage Medical Group Virginia Crosson Cancer Center, Fullerton, California
  - University of California at Los Angeles Dept. of UCLA, Los Angeles, California
  - Ventura County Hematology and Oncology, Oxnard, California
  - Cancer Care Associates Medical Group Dept. of CCA, Redondo Beach, California
  - Santa Barbara Hematolgy Oncology Medical Group Dept.ofSantaBarbaraHem/Onc, Santa Barbara, California
  - Central Coast Medical Oncology Corporation Onc Dept, Santa Maria, California
  - Rocky Mountain Cancer Centers RMCC - Denver-Midtown (3), Greenwood Village, Colorado
  - Florida Cancer Specialists Dept.of FloridaCancerSpec. (2), Fort Myers, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Central Indiana Cancer Centers CICC - East (3), Indianapolis, Indiana
  - Kansas City Cancer Center Dept. of KCCC, Overland Park, Kansas
  - University of Nebraska Medical Center Unv Nebraska Med Ctr (2), Omaha, Nebraska
  - New York Oncology Hematology NYOH Amsterdam, Albany, New York
  - Beth Israel Medical Center Dept.ofBeth Israel Med. Ctr(2), New York, New York
  - Northwest Cancer Specialists Vancouver Cancer Center (3), Portland, Oregon
  - Sarah Cannon Research Institute Dept.ofSarahCannonCancerCtr(5), Nashville, Tennessee
  - Texas Oncology Charles A. Sammons Cancer Ctr, Dallas, Texas
  - Texas Oncology P A SC-Austin, Dallas, Texas
  - Tyler Cancer Center Dept.ofTylerCancerCtr. (2), Tyler, Texas
  - Virginia Oncology Associates SC, Norfolk, Virginia
  - Virginia Cancer Institute VCI (3), Richmond, Virginia
- Argentina (7):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Posadas, Misiones Province
  - Novartis Investigative Site, Rosario, Sante Fe
  - Novartis Investigative Site, Rio Negro, Viedma
  - Novartis Investigative Site, Capital Federal
  - Novartis Investigative Site, Córdoba
- Australia (2):
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, East Bentleigh, Victoria
- Belgium (5):
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Verviers
  - Novartis Investigative Site, Wilrijk
  - Novartis Investigative Site, Yvoir
- Brazil (3):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (2):
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Saint-Jérôme, Quebec
- China (8):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Colombia (4):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Florida Blanca
  - Novartis Investigative Site, Montería
- Egypt (2):
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- France (7):
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Thonon-les-Bains
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Münster
- Greece (4):
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Hong Kong (3):
  - Novartis Investigative Site, Shatin, New Territories, Hong Kong
  - Novartis Investigative Site, Hong Kong SAR
  - Novartis Investigative Site, Tuenmen
- Ireland (2):
  - Novartis Investigative Site, Wilton, Cork
  - Novartis Investigative Site, Dublin
- Italy (5):
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Camposampiero, PD
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Japan (15):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Sakyo-ku, Kyoto
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Kitaadachi-gun, Saitama
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Osaka
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Zaragoza, Veracruz
- Peru (2):
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, Surquillo, Lima region
- San Juan VA Hospital San Juan Hospital, San Juan, Puerto Rico
- Russia (3):
  - Novartis Investigative Site, Kazan', Tatarstan Republic
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- South Africa (3):
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Pretoria
- South Korea (3):
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Switzerland (2):
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Zurich
- Taiwan (5):
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir
- United Kingdom (3):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Sutton
- Novartis Investigative Site, Valencia, Carabobo, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Toi M, Shao Z, Hurvitz S, Tseng LM, Zhang Q, Shen K, Liu D, Feng J, Xu B, Wang X, Lee KS, Ng TY, Ridolfi A, Noel-Baron F, Ringeisen F, Jiang Z. Efficacy and safety of everolimus in combination with trastuzumab and paclitaxel in Asian patients with HER2+ advanced breast cancer in BOLERO-1. Breast Cancer Res. 2017 Apr 11;19(1):47. doi: 10.1186/s13058-017-0839-0. PMID 28399902
- [Derived] Buyse M, Hurvitz SA, Andre F, Jiang Z, Burris HA, Toi M, Eiermann W, Lindsay MA, Slamon D. Statistical controversies in clinical research: statistical significance-too much of a good thing .... Ann Oncol. 2016 May;27(5):760-2. doi: 10.1093/annonc/mdw047. Epub 2016 Feb 9. PMID 26861602
- [Derived] Hurvitz SA, Andre F, Jiang Z, Shao Z, Mano MS, Neciosup SP, Tseng LM, Zhang Q, Shen K, Liu D, Dreosti LM, Burris HA, Toi M, Buyse ME, Cabaribere D, Lindsay MA, Rao S, Pacaud LB, Taran T, Slamon D. Combination of everolimus with trastuzumab plus paclitaxel as first-line treatment for patients with HER2-positive advanced breast cancer (BOLERO-1): a phase 3, randomised, double-blind, multicentre trial. Lancet Oncol. 2015 Jul;16(7):816-29. doi: 10.1016/S1470-2045(15)00051-0. Epub 2015 Jun 16. PMID 26092818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 717 patients were planned to be randomized. A total of 719 patients were randomized between 10-Sep-2009 and 16-Dec-2012.
  Not completed reasons = primary reasons for end of treatment
Period: Overall Study
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Started | 480 | 239
Untreated | 8 | 1
Completed | 0 | 0
Not Completed | 480 | 239
Not completed — Untreated | 8 | 1
Not completed — Adverse Event | 63 | 11
Not completed — Abnormal test procedure result(s) | 1 | 0
Not completed — Disease progression | 259 | 162
Not completed — New cancer therapy | 25 | 7
Not completed — Protocol Violation | 5 | 2
Not completed — Withdrawal by Subject | 66 | 33
Not completed — Lost to Follow-up | 2 | 0
Not completed — Administrative problems | 39 | 23
Not completed — Death | 12 | 0

BASELINE CHARACTERISTICS:
Population: The FAS consisted of all randomized patients. Following the intent-to-treat principle patients were analyzed according to the treatment and stratum they were assigned to at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab | Total
Number analyzed (Participants) | 480 | 239 | 719
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (11.46) | 52.1 (11.63) | 53.0 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 480 | 239 | 719
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 214 | 97 | 311
  Black | 26 | 12 | 38
  Asian | 198 | 105 | 303
  Native American | 3 | 0 | 3
  Other | 39 | 25 | 64

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Investigators' Assessment Based on Local Radiology Review - Full Population
Description: PFS is defined as the time from the date of randomization to the date of first documented tumor progression or death from any cause, whichever occurs first. This was assessed in the full patient population.
Time Frame: date of randomization to the date of first documented tumor progression or death from any cause, whichever occurs first, reported between day of first patient randomized up to about 56 months
Population: The Full Analysis Set (FAS) consists of all randomized patients. Following the intent-to-treat principle patients will be analyzed according to the treatment and stratum they were assigned to at randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 480 | 239
months | 14.95 [14.55 to 17.91] | 14.49 [12.29 to 17.08]
Statistical Analysis 1: Comparison: Everolimus + Paclitaxel + Trastuzumab vs Placebo + Paclitaxel + Trastuzumab; Test type: Superiority; p = 0.1166, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.73 to 1.08]

2. Primary Outcome: Progression-free Survival (PFS) Per Investigators' Assessment Based on Local Radiology Review - (Hormone Receptor (HR)-Negative Population
Description: PFS is defined as the time from the date of randomization to the date of first documented tumor progression or death from any cause, whichever occurs first. This was assessed in the HR-negative patient population.
Time Frame: as for outcome 1
Population: HR-negative Full Analysis Set (HR-negative FAS) consists of subset of patients from the FAS population with HR-negative status at Baseline.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 208 | 103
Months | 20.27 [14.95 to 24.08] | 13.08 [10.05 to 16.56]
Statistical Analysis 1: Comparison: Everolimus + Paclitaxel + Trastuzumab vs Placebo + Paclitaxel + Trastuzumab; Test type: Superiority; p = 0.0049, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.48 to 0.91]

3. Secondary Outcome: Overall Survival (OS) - Full Population
Description: OS is defined as the time from date of randomization to the date of death due to any cause. For patients with documented progression, survival follow up was performed either by telephone or clinic visit at least every 3 months. Additional survival updates were requested prior to interim or final analysis or prior to providing data to the health authorities. This was assessed in the full patient population.
Time Frame: up to about 76 months
Population: The Full Analysis Set (FAS) consists of all randomized patients. Following the intent-to-treat principle patients will be analyzed according to the treatment and stratum they were assigned to at randomization. Due to the exploratory nature of the OS analysis, OS was not statistically tested
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 480 | 239
Months | 48.56 [40.94 to 58.94] | 49.97 [40.84 to NA] — N/A = The upper limit of the Confidence Interval was not estimable as there were not enough events.

4. Secondary Outcome: Overall Survival (OS) - HR-negative Population
Description: OS is defined as the time from date of randomization to the date of death due to any cause. For patients with documented progression, survival follow up was performed either by telephone or clinic visit at least every 3 months. Additional survival updates were requested prior to interim or final analysis or prior to providing data to the health authorities. This was assessed in the HR-negative patient population.
Time Frame: up to about 76 months
Population: HR-negative Full Analysis Set (HR-negative FAS) consists of subset of patients from the FAS population with HR-negative status at Baseline. Due to the exploratory nature of the OS analysis, OS was not statistically tested.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 208 | 103
Months | 56.97 [44.09 to NA] — N/A = The upper limit of the Confidence Interval was not estimable as there were not enough events. | 41.63 [34.83 to NA] — N/A = The upper limit of the Confidence Interval was not estimable as there were not enough events.

5. Secondary Outcome: Overall Response Rate (ORR) - Full Population
Description: ORR is defined as the percentage of participants whose best overall response is either complete response (CR) or partial response (PR) according to RECIST. This was assessed in the full patient population. Complete response is achieved when all lesions evaluated at Baseline are absent at subsequent visit.
Time Frame: up to about 23 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 480 | 239
Percentage of participants | 67.1 [62.7 to 71.3] | 69.0 [62.8 to 74.8]
Statistical Analysis 1: Comparison: Everolimus + Paclitaxel + Trastuzumab vs Placebo + Paclitaxel + Trastuzumab; Test type: Superiority; p = 0.7276, Exact Cochran-Mantel-Haenzel chi-square

6. Secondary Outcome: Overall Response Rate (ORR) - HR-negative Population
Description: ORR is defined as the percentage of participants whose best overall response is either complete response (CR) or partial response (PR) according to RECIST. This was assessed in a subset of patients with Hormone Receptor Negative disease. Complete response is achieved when all lesions evaluated at Baseline are absent at subsequent visit.
Time Frame: up to about 23 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 208 | 103
Percentage of participants | 73.1 [66.5 to 79.0] | 70.9 [61.1 to 79.4]
Statistical Analysis 1: Comparison: Everolimus + Paclitaxel + Trastuzumab vs Placebo + Paclitaxel + Trastuzumab; Test type: Superiority; p = 0.4085, Exact Cochran-Mantel-Haenzel chi-square

7. Secondary Outcome: Clinical Benefit Rate (CBR) Equal to or Greater Than 24 Weeks - Full Population
Description: CBR is defined as the percentage of participants whose best overall response is either complete response (CR), a partial response (PR) or stable disease (SD) lasting for at least 24 weeks, according to RECIST. This was assessed in the full patient population. Complete response is achieved when all lesions evaluated at Baseline are absent at subsequent visit.
Time Frame: up to about 23 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 480 | 239
Percentage of participants | 75.8 [71.7 to 79.6] | 81.2 [75.6 to 85.9]
Statistical Analysis 1: Comparison: Everolimus + Paclitaxel + Trastuzumab vs Placebo + Paclitaxel + Trastuzumab; Test type: Superiority; p = 0.9573, Exact Cochran-Mantel-Haenzel chi-square

8. Secondary Outcome: Clinical Benefit Rate (CBR) Equal to or Greater Than 24 Weeks - HR-negative Population
Description: CBR is defined as the percentage of participants whose best overall response is either complete response (CR), a partial response (PR) or stable disease (SD) lasting for at least 24 weeks, according to RECIST. This was assessed in a subset of patients with Hormone Receptor Negative disease. Complete response is achieved when all lesions evaluated at Baseline are absent at subsequent visit.
Time Frame: up to about 23 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 208 | 103
Percentage of participants | 78.8 [72.7 to 84.2] | 79.6 [70.5 to 86.9]
Statistical Analysis 1: Comparison: Everolimus + Paclitaxel + Trastuzumab vs Placebo + Paclitaxel + Trastuzumab; Test type: Superiority; p = 0.6382, Exact Cochran-Mantel-Haenzel chi-square

9. Secondary Outcome: Time to Overall Response Based on Investigator - Full Population
Description: Time to overall response defined as the time between date of randomization until first documented response Complete reseponse (CR) or partial response (PR) ), according to RECIST. This was assessed in the full patient population and in a subset of patients with Hormone Receptor Negative disease. Complete response is achieved when all lesions evaluated at Baseline are absent at subsequent visit.
Time Frame: up to about 23 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 480 | 239
months | 2.10 [2.00 to 3.58] | 2.00 [1.94 to 2.27]

10. Secondary Outcome: Time to Overall Response Based on Investigator - HR-negative Population
Description: as for outcome 9
Time Frame: up to about 23 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 208 | 103
months | 1.94 [1.87 to 2.00] | 1.97 [1.87 to 3.58]

11. Secondary Outcome: Overall Response (OR) - Full Population
Description: OR applies only to patients whose best OR was CR or PR. Start date = date of first documented response (CR or PR) and end date = date of documented response (CR or PR) and end date = date of event defined as the first documented progression or death due to underlying cause. Complete response is achieved when all lesions evaluated at Baseline are absent at subsequent visit.
Time Frame: up to about 23 months
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 480 | 239
Percentage of participants
  Complete Response (CR) | 5.6 | 5.9
  Partial Response (PR) | 61.5 | 63.2

12. Secondary Outcome: Overall Response (OR) - HR-negative Population
Description: OR applies only to patients whose best OR was CR or PR. Start date = date of first documented response (CR or PR) and end date = date of documented response (CR or PR) and end date = date of event defined as the first documented progression or death due to underlying cause. This was assessed in the HR-negative patient population. Complete response is achieved when all lesions evaluated at Baseline are absent at subsequent visit.
Time Frame: up to about 23 months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 208 | 103
Percentage of participants
  Complete Response (CR) | 7.7 | 2.9
  Partial Response (PR) | 65.4 | 68.0

13. Secondary Outcome: Everolimus Blood Level Concentrations at Steady States for Everolimus
Description: Blood levels at steady states for everolimus 10 mg/day and 5 mg/day. Only valid samples are included. Some patients had dose reduction to 5 mg daily dose therefore the everolimus blood concentration for them have been summarized separately. Cycle = 28 days
Time Frame: predose, 2 hours post-dose at Cycle 2/Day 1, Cycle 2/Day 15, Cycle 2/ Day 22
Population: Safety Set: consists of all patients who received at least 1 dose of study treatment & have at least 1 valid post-baseline safety assessment. Patients were analyzed according to the treatment actually received. If patient took at least 1 dose of treatment to which he/she was randomized then the treatment actually received was the rand. treatment.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Everolimus 10 mg/Day: Everolimus 10 mg daily
- Everolimus 5 mg/Day: Everolimus 5 mg daily
Arm/Group | Everolimus 10 mg/Day | Everolimus 5 mg/Day
Number analyzed (Participants) | 60 | 21
ng/mL
  Pre-dose (Cmin) @ C2D1: number analyzed (Participants) | 54 | 14
  Pre-dose (Cmin) @ C2D1 | 14.380 (10.0169) | 7.959 (8.1546)
  2 hrs post administration (C2h) @ C2D1: number analyzed (Participants) | 60 | 17
  2 hrs post administration (C2h) @ C2D1 | 44.485 (22.1986) | 23.449 (10.4112)
  Pre-dose (Cmin) @ C2D15: number analyzed (Participants) | 44 | 17
  Pre-dose (Cmin) @ C2D15 | 13.206 (9.9821) | 5.473 (3.9690)
  2 hrs post administration (C2h) @ C2D15: number analyzed (Participants) | 44 | 21
  2 hrs post administration (C2h) @ C2D15 | 43.494 (21.5940) | 20.329 (7.9518)
  Pre-dose (Cmin) @ C2D22: number analyzed (Participants) | 40 | 17
  Pre-dose (Cmin) @ C2D22 | 13.432 (13.2782) | 7.494 (5.8503)
  2 hrs post administration (C2h) @ C2D22: number analyzed (Participants) | 48 | 21
  2 hrs post administration (C2h) @ C2D22 | 43.947 (28.0107) | 22.192 (10.9277)

14. Secondary Outcome: Paclitaxel Plasma Concentrations
Description: Blood levels at steady states for everolimus/placebo
Time Frame: Cycle 2/Day 15 (Pre-infusion and end of infusion)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Everolimus: Everolimus 10 mg/day
- Everolimus Placebo: Placebo of everolimus 10 mg daily
Arm/Group | Everolimus | Everolimus Placebo
Number analyzed (Participants) | 91 | 43
ng/mL
  Pre-infusion (Cmin) @ C2D15 | 1.424 (5.8645) | 0 (0)
  End of infusion (Cmax) @ C2D15: number analyzed (Participants) | 65 | 33
  End of infusion (Cmax) @ C2D15 | 5159.338 (15473.636) | 4296.697 (7431.0799)

15. Secondary Outcome: Trastuzumab Serum Concentrations
Description: Blood levels at steady states for everolimus/placebo
Time Frame: Cycle 4/Day 1 (Pre-infusion and end of infusion)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: microgram/ml
Groups:
- Everolimus + Trastuzumab: Everolimus plus trastuzumab
Arm/Group | Everolimus + Trastuzumab | Everolimus Placebo
Number analyzed (Participants) | 98 | 54
microgram/ml
  Pre-infusion (Cmin) @ C4D1 | 26.606 (9.6548) | 29.180 (12.1252)
  End of infusion (Cmax) @ C4D1: number analyzed (Participants) | 83 | 46
  End of infusion (Cmax) @ C4D1 | 64.296 (23.4635) | 67.643 (20.8852)

16. Secondary Outcome: Time to Deterioration of Eastern Cooperative Oncology Group Performance Status (ECOG-PS) Score - Full Population
Description: Time to definitive deterioration of the ECOG PS by one category of the score from baseline will be performed. Baseline is the last available assessment on or before randomization date. A deterioration is considered definitive if no improvements in the ECOG PS status is observed at a subsequent time of measurement during the treatment period following the time point where the deterioration is observed.
Time Frame: up to about 56 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 480 | 239
months | 39.20 [31.31 to NA] — N/A = not enough number of events in a treatment arm, so the upper limit of 95% CI was not reached and hence data was presented as N/A | NA [30.39 to NA] — N/A = not enough number of events in a treatment arm, so the median was not reached and hence data was presented as N/A

17. Secondary Outcome: Time to Deterioration of Eastern Cooperative Oncology Group Performance Status (ECOG-PS) Score - HR-negative Population
Description: as for outcome 16
Time Frame: up to about 56 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Paclitaxel + Trastuzumab | Placebo + Paclitaxel + Trastuzumab
Number analyzed (Participants) | 208 | 103
months | NA [25.56 to NA] — N/A = not enough number of events in a treatment arm, so the median and upper limit of 95% CI were not reached and hence data was presented as N/A | NA [26.91 to NA] — N/A = not enough number of events in a treatment arm, so the median and upper limit of 95% CI were not reached and hence data was presented as N/A

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Patient First Treatment until 30 days after Last Patient Last Visit.
Groups:
- Everolimus+ Paclitaxel+ Trastuzumab: Everolimus 10 mg daily in combination with paclitaxel 80mg/m2 weekly on days 1, 8, 15 and trastuzumab 2mg/kg weekly on days 1, 8, 15, 22
- Placebo+ Paclitaxel+ Trastuzumab: Placebo of everolimus 10 mg daily in combination with paclitaxel 80mg/m2 weekly on days 1, 8, 15 and trastuzumab 2mg/kg weekly on days 1, 8, 15, 22
Arm/Group | Everolimus+ Paclitaxel+ Trastuzumab | Placebo+ Paclitaxel+ Trastuzumab
All-Cause Mortality (participants affected / at risk) | 23/472 | 2/238
Serious Adverse Events (participants affected / at risk) | 173/472 | 40/238
Other Adverse Events (participants affected / at risk) | 466/472 | 236/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus+ Paclitaxel+ Trastuzumab (N=472) | Placebo+ Paclitaxel+ Trastuzumab (N=238)
Anaemia (Blood and lymphatic system disorders) | 6 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Cataract (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 2 | 0
Ocular surface disease (Eye disorders) | 1 | 0
Strabismus (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 10 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 1 | 0
Calcinosis (General disorders) | 0 | 1
Catheter site related reaction (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 12 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Breast abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 5 | 4
Clostridium colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 10 | 2
Fungal infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 2 | 0
Mastitis (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 22 | 0
Pneumonia klebsiella (Infections and infestations) | 2 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Pulmonary tuberculoma (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Salmonellosis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 1
Septic shock (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 7 | 0
Urosepsis (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3
Injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood potassium decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 0
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 3
Ataxia (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 2
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Thrombosis in device (Product Issues) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 1
Conversion disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1
Breast ulceration (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 21 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus+ Paclitaxel+ Trastuzumab (N=472) | Placebo+ Paclitaxel+ Trastuzumab (N=238)
Anaemia (Blood and lymphatic system disorders) | 143 | 38
Leukopenia (Blood and lymphatic system disorders) | 71 | 24
Neutropenia (Blood and lymphatic system disorders) | 177 | 59
Thrombocytopenia (Blood and lymphatic system disorders) | 46 | 6
Left ventricular dysfunction (Cardiac disorders) | 32 | 10
Abdominal pain (Gastrointestinal disorders) | 71 | 29
Abdominal pain upper (Gastrointestinal disorders) | 55 | 26
Aphthous ulcer (Gastrointestinal disorders) | 25 | 4
Constipation (Gastrointestinal disorders) | 101 | 51
Diarrhoea (Gastrointestinal disorders) | 267 | 112
Dyspepsia (Gastrointestinal disorders) | 50 | 26
Haemorrhoids (Gastrointestinal disorders) | 32 | 7
Mouth ulceration (Gastrointestinal disorders) | 60 | 14
Nausea (Gastrointestinal disorders) | 154 | 83
Stomatitis (Gastrointestinal disorders) | 315 | 77
Toothache (Gastrointestinal disorders) | 35 | 21
Vomiting (Gastrointestinal disorders) | 122 | 55
Asthenia (General disorders) | 94 | 41
Chills (General disorders) | 29 | 6
Fatigue (General disorders) | 168 | 87
Oedema peripheral (General disorders) | 156 | 59
Pain (General disorders) | 28 | 12
Peripheral swelling (General disorders) | 30 | 10
Pyrexia (General disorders) | 181 | 63
Cellulitis (Infections and infestations) | 28 | 8
Influenza (Infections and infestations) | 36 | 24
Nasopharyngitis (Infections and infestations) | 90 | 47
Paronychia (Infections and infestations) | 26 | 8
Pharyngitis (Infections and infestations) | 25 | 5
Pneumonia (Infections and infestations) | 33 | 10
Rhinitis (Infections and infestations) | 30 | 14
Upper respiratory tract infection (Infections and infestations) | 67 | 34
Urinary tract infection (Infections and infestations) | 56 | 17
Alanine aminotransferase increased (Investigations) | 95 | 45
Aspartate aminotransferase increased (Investigations) | 72 | 29
Ejection fraction decreased (Investigations) | 35 | 15
Haemoglobin decreased (Investigations) | 41 | 8
Neutrophil count decreased (Investigations) | 44 | 23
Weight decreased (Investigations) | 99 | 13
Weight increased (Investigations) | 19 | 26
White blood cell count decreased (Investigations) | 34 | 14
Decreased appetite (Metabolism and nutrition disorders) | 110 | 36
Hypercholesterolaemia (Metabolism and nutrition disorders) | 88 | 23
Hyperglycaemia (Metabolism and nutrition disorders) | 58 | 13
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 68 | 17
Hypocalcaemia (Metabolism and nutrition disorders) | 24 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 68 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 80 | 41
Back pain (Musculoskeletal and connective tissue disorders) | 72 | 42
Bone pain (Musculoskeletal and connective tissue disorders) | 30 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 33 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 37 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 78 | 45
Pain in extremity (Musculoskeletal and connective tissue disorders) | 86 | 39
Dizziness (Nervous system disorders) | 74 | 37
Dysgeusia (Nervous system disorders) | 59 | 24
Headache (Nervous system disorders) | 130 | 70
Hypoaesthesia (Nervous system disorders) | 61 | 36
Neuropathy peripheral (Nervous system disorders) | 136 | 58
Neurotoxicity (Nervous system disorders) | 40 | 24
Paraesthesia (Nervous system disorders) | 35 | 25
Peripheral sensory neuropathy (Nervous system disorders) | 61 | 37
Anxiety (Psychiatric disorders) | 31 | 12
Depression (Psychiatric disorders) | 23 | 12
Insomnia (Psychiatric disorders) | 78 | 39
Dysuria (Renal and urinary disorders) | 40 | 9
Breast pain (Reproductive system and breast disorders) | 26 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 191 | 80
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 22 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 110 | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 156 | 43
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 74 | 31
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 66 | 11
Productive cough (Respiratory, thoracic and mediastinal disorders) | 25 | 14
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 43 | 18
Acne (Skin and subcutaneous tissue disorders) | 29 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 221 | 125
Dry skin (Skin and subcutaneous tissue disorders) | 37 | 20
Erythema (Skin and subcutaneous tissue disorders) | 49 | 16
Nail disorder (Skin and subcutaneous tissue disorders) | 68 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 64 | 24
Rash (Skin and subcutaneous tissue disorders) | 191 | 49
Hot flush (Vascular disorders) | 13 | 12
Hypertension (Vascular disorders) | 74 | 27

LIMITATIONS AND CAVEATS:
Of the 480 patients enrolled in the Everolimus arm, 8 were untreated and in the Placebo arm, of the 239 patients enrolled, 1 was untreated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.